CLINICAL TRIAL: NCT04725825
Title: Central Pain Modulatory Effects of Dry-Needling in Patients With Non-Specific Neck Pain: a Randomized Controlled Experimental Study
Brief Title: Central Pain Modulatory Effects of Dry-Needling in Patients With Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Principal Investigator, VakgroepRevalidatiewetenschappen, Principal Investigator, University Ghent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BC-05419
Record Dates: First submitted 2020-09-24; First posted 2021-01-27 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Neck Pain, Posterior; Trapezius Muscle Strain
Keywords: Dry Needling; Sham Needling; Myofascial Pain Syndrome; Central Pain Modulatory Effects
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): A single dry needling session will be performed on the dominant painful trapezius muscle, with the patient lying in prone position. After palpation of a taut band, and detection of a MTrP in the upper trapezius muscle, a trained physiotherapist will penetrate the needle into skin surface, fascia, into the muscle tissue at the MTrP location, and will move the needle up and down (fast-in, fast-out technique) in three different directions.
  In case local twitch responses are elicited, this will be repeated until the local twitch responses are extinct.
  Interventions: Other: Dry needling
- Sham needling (Sham Comparator): A single sham needling session will be performed with the subject lying on the non painful side. After palpation of a taut band, and detection of a MTrP in the upper trapezius muscle, a trained physiotherapist will penetrate the needle into the skin surface at the MTrP location. The fascia and muscle tissue will not be penetrated.
  Interventions: Other: Sham needling

INTERVENTIONS:
Other: Dry needling — Dry needling (DN) is a myofascial treatment technique, in which a thin, solid filiform needle is inserted directly into the MTrP. During dry needling, local twitch responses (LTR) can be elicited. These are involuntary contractions of muscle fibers, leading to muscle relaxation, an increase in blood flow,recovery of the muscle metabolism and thus a reduction of pain and stiffness.
  Arms: Dry needling
Other: Sham needling — During sham needling, a solid, filiform needle is inserted in the skin surface at the trigger point location, without penetrating the fascia and muscle tissue.
  Arms: Sham needling

SUMMARY:
An experimental study will be conducted to evaluate the effect of a single dry needling session, compared to a sham needling session, on pain intensity, local and peripheral hyperalgesia, and conditioned pain modulation in patients with chronic idiopathic neck pain.

DETAILED DESCRIPTION:
Chronic idiopathic neck pain frequently has a myofascial origin. This cervical myofascial pain is caused by myofascial trigger points (MTrPs). Myofascial trigger points are defined as hyperirritable nodules in a contracture of skeletal muscle fibers, which can cause pain symptoms, motor symptoms as well as autonomic symptoms.

Many chronic pain populations (e.g. chronic whiplash associated disorders, fibromyalgia, chronic low back pain) show impaired pain processing and signs of central sensitisation. Central pain processing is defined as an increased responsivity of the nociceptive neurons in the central nerve system and is characterized by hyperalgesia (increased pain after a painful stimuli), allodynia (pain caused by a non-painful stimuli) and temporal summation (increased pain response after repeated stimuli with the same intensity). Hyperalgesia can be divided in local (increased sensitivity in the area of the complaints) and peripheral (increased sensitivity at remote area's). Furthermore, deficient inhibitory pain modulation can be present in this population. Conditioned pain modulation (CPM) can be measured by combining a painful conditioning stimuli (e.g. cold or heat) on a remote location, with a painful test stimuli.

Cervical myofascial pain is often treated by dry needling (DN). DN is a myofascial treatment technique, which has been gaining interest in recent years. During DN, a thin, solid filiform needle is inserted directly into the MTrP. During this treatment, local twitch responses can be elicited. These are involuntary contractions of muscle fibers, leading to muscle relaxation, an increased local blood flow, recovery of the muscle metabolism and thus a reduction of pain and stiffness. By deactivation of the source of pain, chronification of the pain can be prevented.

Up to this moment, there are no studies that investigated the central effects of DN. The aim of this study is to compare the effects of DN with sham needling on pain intensity, local and peripheral hyperalgesia and CPM, in patients with chronic idiopathic neck pain. Therefore, 100 patients will be recruited. Participants are included based on online questionnaires, a clinical examination of neck and shoulder, and the identification of a MTrP in the upper trapezius muscle. All participants will receive information and have to sign an informed consent form. Participants will be subjected to baseline assessment, which involves measurements of pain scores, hyperalgesia (pressure pain thresholds (PPT) by algometry) and CPM (by combining immersion of the hand in hot water while repeating the PPT). Then, participants will be randomly allocated to either a dry needling group or a sham needling group. The dry needling group will receive a dry needling treatment at the identified trigger point location of the upper trapezius, whereas the sham needling group will receive an intervention in which the needle only penetrates the skin but not the fascia and muscle tissue. The one-time intervention of both groups will take approximately 15 minutes. After the treatment, the baseline measurements will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain (symptom duration >3 months)
* Mean NRS score >3/10
* The presentation of a clinically relevant myofascial triggerpoint in the upper trapezius muscle.

Exclusion Criteria:

* Specific neck pain (eg.structural pathology like a cervical discus hernia, cervical nerve root compression, factures...)
* Major depression or psychiatric illness
* Cardiovascular, neurological, life threatening, systemic and metabolic diseases
* Other transferable diseases (HIV, hepatitis...)
* Coagulation disorders or use of coagulation medication
* Pregnancy or given birth the last year
* Traumatic injuries/surgery to neck and upper limb region
* Diagnosis of fibromyalgia/chronic fatigue syndrome
* BMI > 30 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change in distant Pressure Pain Threshold | Baseline and immediately after the intervention
  A distant standardised PPT will be assessed using a digital handheld pressure algometer (FDX; Wagner Instruments) at the quadriceps muscle of the dominant painful side to measure distant hyperalgesia.
  To measure the PPT, the researcher will apply the digital algometer to each of the indicated points with a round rubber end of 1 cm² and an increasing pressure of circa 1 N/s. As soon as the sensation of the subject shifts from a comfortable pressure to an altered, unpleasant feeling, the participant reports this and the test will be finished.
  Each point will be measured twice with a 30-second interval in between and all measurements will be performed by one researcher in the same standardised position for each point and will be executed in a randomised order per patient.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | Baseline and immediately after the intervention
  The neck pain of the patients will be rated on an 11-point NRS at the beginning of the trial. After the hot water immersion (CPM; at baseline and post-intervention), patients will also be asked to score the pain caused by the hot water on a NRS. Minimum value is zero; a score of zero means no pain (= better outcome) and maximum score is 10, which indicates the worst pain possible (=worse outcome).
Change in Conditioned Pain Modulation | baseline and immediately after the intervention
  Participants will be asked to put their (non-dominant) hand (up to a marked line on the wrist) in a bath (VersaCool, Thermo Fisher Scientific, Waltham, Massachusetts) with demineralised circulating water maintained at 46,5°C for one minute. To maximise the CPM effect, the non-dominant hand will be used.
  During this minute, participants will be encouraged to persevere after 30 and after 45 seconds by one of the investigators. The PPTs will be used as the test stimulus.These will be measured pre- and post immersion.The difference between the pre- and post immersion PPTs will be used to assess the effectiveness of the CPM.
Change in local Pressure Pain Threshold | Baseline and immediately after the intervention
  Two local standardised PPTs will be assessed using a digital handheld pressure algometer (FDX; Wagner Instruments) at the dominant painful and non-dominant painful upper trapezius muscle to measure local hyperalgesia.
  To measure the PPT, the researcher will apply the digital algometer to each of the indicated points with a round rubber end of 1 cm² and an increasing pressure of circa 1 N/s. As soon as the sensation of the subject shifts from a comfortable pressure to an altered, unpleasant feeling, the participant reports this and the test will be finished.
  Each point will be measured twice with a 30-second interval in between and all measurements will be performed by one researcher in the same standardised position for each point and will be executed in a randomised order per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Meeus, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No